CLINICAL TRIAL: NCT02389218
Title: A Prospective Study of Medical Therapy Against Cryoballoon Ablation in Symptomatic Recent Onset Persistent Atrial Fibrilation
Brief Title: A Prospective Study of Medical Therapy Against Cryoballoon Ablation in Symptomatic Recent Onset Persistent AF
Acronym: METACSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/1113
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cryoablation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone; Sotalol; Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryoablation (Experimental): Cryoballoon single ablation (as described in the reference) at entry after randomization to this group. Single procedure,not to be repeated.
  Interventions: Device: single ablation (CryoBalloonAblation (CBA)
- Drug (Active Comparator): Conventional, available anti arrhythmic drugs (propafenone, sotalol or flecainide), in a first stage, sequential, with amiodarone in second stage
  Interventions: Drug: sequential drug adjustment (propafenone, sotalol or flecainide)

INTERVENTIONS:
Device: single ablation (CryoBalloonAblation (CBA) — Cryoablation at entry, after randomization to this group
  Arms: Cryoablation
Drug: sequential drug adjustment (propafenone, sotalol or flecainide) — Correct drug dosage at entry, sequential adjustment / titration, in stage 2 amiodarone
  Arms: Drug

SUMMARY:
Prospective trial comparing the efficacy and safety of CryoBalloonAblation (CBA) to standardized medication for treatment of early onset persistent atrial fibrillation (AF) without structural heart disease. The value of CBA in these patients has never been studied; the endpoints for persistent patients are much easier than for paroxysmal patients. Reduction in left atrial (LA) size will be compared versus patients on drug therapy and versus failing patients.

DETAILED DESCRIPTION:
The total AF history should be shorter than 24 months. Symptomatic patients can be included if they have had within the last year at least 2 episodes of documented AF, lasting minimal 30 sec. One episode in the entire history should have lasted more than 48 h, requiring electrical or pharmacological cardioversion or stopped spontaneously after more than 7 days.

All patients eligible for the study will sign informed consent, have an echocardiogram prior to inclusion to exclude severe left ventricular dysfunction, to rule out significant valve abnormalities, left ventricular hypertrophy and to assess the LA volume and diameter.

Prior to randomization, and after inclusion it is suggested to the local investigators to perform an MRI-scan or CT scan of the LA and pulmonary veins (in both branches of the study ) in eligible patients to assess the anatomy and the left atrial volume. The results should not influence the strategy of treatment.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years and legally capable
* First documentation or history of symptomatic AF more than 30 sec within the last 2 years
* Twice AF within the last year
* One episode cardioverted after more than 48 hours or spontaneously terminated after more than 7 days
* Eligible for at least one first step drug therapy (sotalol, propafenone, or flecainide) and for amiodarone
* Left ventricular ejection fraction estimated > 45%
* LA diameter < 50 mm (parasternal short axis) and LA volume less than 100 ml (apical view, Area Length method;)
* CHADS2 ≤ 2
* Failed AAD strategy, or untreated with AAD
* No use of Amiodarone in the previous 3 months (except IV or oral for 7 days)
* Informed consent

Exclusion Criteria:

* Age > 75 yrs
* CHF
* Ischemic heart disease as known in the history
* (Severe) Left ventricular hypertrophy as shown on echo (IVSd or PWd > 14 mm)
* Hyperthyroidism
* Congenital heart disease
* Hypertrophic Cardiomyopathy, Arrhythmogenic Right ventricular Cardiomyopathy, channelopathies
* Contra-indications to AAD
* Long QT syndrome
* Received already adequately dosed all level 1 drugs (sotalol, propafenone, and flecainide)
* Pure (typical) atrial flutter as documented on one occasion

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Sinus rhythm | one year
  Sinus rhythm at one year

SECONDARY OUTCOMES:
Reduction LA volume | one year
  Reduction left atrial volume in successfully treated patients
Number of cardioversions | one year
  Number of cardioversions
Percentage on anti arrhythmic drugs (AAD) | 6 months
  Percentage on AAD in each group
Percentage on AAD | 12 months
  Percentage on AAD in each group
Vascular complications | one year
  Vascular complications, including tamponade
Stroke, transient ischemic attack (TIA) | one year
  Stroke, TIA (symptomatic)
Serious adverse events (SAE) | one year
  Adverse events leading to admission or death
Freedom of AF | one year
  Freedom of atrial fibrillation with all means

CONTACTS AND LOCATIONS:
Overall Officials: Luc Jordaens, MD, PhD, Principal Investigator — Professor of Cardiology
Locations (3):
- Belgium (3):
  - Brussels Heart Centre, Brussels
  - Saint Luc, Brussels
  - Dept Cardiologie, Ghent

REFERENCES:
- [Background] Van Belle Y, Janse P, Theuns D, Szili-Torok T, Jordaens L. One year follow-up after cryoballoon isolation of the pulmonary veins in patients with paroxysmal atrial fibrillation. Europace. 2008 Nov;10(11):1271-6. doi: 10.1093/europace/eun218. PMID 18955409

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02389218/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02389218/SAP_001.pdf